CLINICAL TRIAL: NCT02672124
Title: A New Micro Swim-up Procedure for Sperm Preparation in ICSI Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cervesi Hospital, Cattolica, Italy (Other)
Responsible Party: Principal Investigator, Palini Simone, Embryologist, Cervesi Hospital, Cattolica, Italy
Other Study IDs: NEW MICRO SWIM-UP PROCEDURE
Record Dates: First submitted 2016-01-19; First posted 2016-02-03 (Estimated); Last update posted 2021-02-09 (Actual); Status verified 2020-02

CONDITIONS: Microswimup Procedure Efficacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The aim of this study is to evaluate the microbiological safety and the efficacy of a new not expensive, easy and fast technique (Direct Microswimup) for sperm preparation in In Vitro Fertilization (IVF) treatments without the use of centrifuge, able to simplify the procedure and to avoid mismatches by ensuring the same results of the standard techniques in terms of fertilization rate, blastulation rate, pregnancy/abortion rate, cryostorage rate, and a better euploid status of the embryos.

ELIGIBILITY:
Inclusion Criteria:

* at least 8 oocytes retrieved at pickup
* oocyte insemination with ICSI technique
* only elective single embryo transfer (eSET) at blastocyst stage
* sperm concentration ≥ 1 X 106 /ml
* absence of antibiotic treatment in the previous four weeks for male patients

Exclusion Criteria:

* recurrent miscarriages
* more than three in vitro fertilization treatment
* azoospermia

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study included couples submitted to in vitro fertilization treatment at the Unit of Physiopathology of Reproduction (Cervesi Hospital, Cattolica, RN, Italy).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
microbiological test | 3 months
  A standard bacteriological culture [based on inoculation of blood and "chocolate" agar plates and Brain-Heart Infusion broth, followed by incubation at 37°C for up to 72 hours] was performed in order to investigate the presence and amount of colonizing bacteria delivered with the semen at ejaculation and after treatment

SECONDARY OUTCOMES:
semen treatment efficacy | 6 months
  number of obtain blastocysts (%) and number of pregnancy (%)

OTHER OUTCOMES:
euploid status | 6 months
  molecular analysis of blastocyst's biopsy

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Cervesi Hospital IVF Unit, Cattolica, Rimini
  - Primiterra Mariangela, Cattolica, Rimini